CLINICAL TRIAL: NCT04490356
Title: A Novel Telehealth Intervention Using Nutrition and Exercise to Extend Intervention Benefits: Enhancing Physical Function in the Long-term for Obese Older Adults
Brief Title: Enhancing Physical Function in the Long-term for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRO00105630; 1P30AG064201-01 (NIH)
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-03

CONDITIONS: Weight Loss Maintenance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Legacy Intervention (Experimental): Older adults who have successfully completed a lifestyle intervention (lost at least 3% body weight and increased short physical performance battery (SPPB) score by 1 point or 6-minute walk test (6MWT) by 50 meters) will be enrolled in a tele-nutrition and tele-exercise intervention.
  Interventions: Behavioral: Legacy Intervention

INTERVENTIONS:
Behavioral: Legacy Intervention — The Legacy intervention is a nutrition and exercise protocol delivered using video conference technology. The Legacy protocol incorporates behavioral strategies along with nutrition and exercise to maintain and extend functional benefits of obesity treatment.

SUMMARY:
The intervention being studied is a 12-week nutrition and physical activity intervention, delivered using videoconference technology by registered dietitian clinicians to maintain weight loss and functional gains in older adults who successfully completed a weight loss intervention. The "Legacy Intervention" will include cognitive behavioral strategies (e.g., goal setting, self-monitoring, and social support), and draw upon a toolbox of e-approaches, including daily and weekly text reminders, virtual exercise classes, virtual individual and group nutrition classes, and step tracking device.

ELIGIBILITY:
Inclusion Criteria:

* Participated in a weight loss intervention in the last 9 months and lost ≥ 3% body weight and improved SPPB score by ≥ 1 point or 6MWT by ≥ 50 meters
* Age ≥ 60
* Able to speak and understand spoken and written English.
* Able to record dietary intake and weight

Exclusion Criteria:

* Presence of unstable or symptomatic life-threatening illness
* Neurological conditions causing functional impairment, including Parkinson's disease, multiple sclerosis, and permanent disability due to stroke
* Inability to complete physical function assessment
* No access to internet connection to participate in the tele-intervention
* Unable or unwilling to use provided tablet to participant in tele-intervention
* History of cognitive impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Starr, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, School of Medicine, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Legacy Intervention
Started | 14
Completed | 13
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Proportion Retention
Description: Proportion retention will be computed by dividing the number of retained subjects at the end of the intervention by the total number of participants
Time Frame: 12 week endpoint
Population: Participants who completed the study
Measure: Number; unit: percent of participants
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 13
percent of participants | 93

2. Primary Outcome: Acceptability as Measured by Participant Satisfaction
Description: Participants will asked to rate their satisfaction by answering the question "Overall, I'm glad I participated in this weight maintenance program" with the following possible responses: 1- strongly disagree , 2- disagree, 3 - neither agree nor disagree, 4- agree, and and 5 -strongly agree. Score ranges from 1- 5 with higher score indicating greater satisfaction
Time Frame: 12 week endpoint
Population: Participants who completed the study; data were not collected for one participant who completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 12
score on a scale | 4.8 (0.4)

3. Secondary Outcome: Change in Physical Performance as Measured by the Short Physical Performance Battery
Description: Scores range from 0 to 12 with higher score indicating better performance.
Time Frame: 0 weeks, 12 weeks
Population: Participants who completed the study; data were not collected for one participant who completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 12
score on a scale
  0 weeks (baseline) | 10.6 (1.2)
  12 weeks | 11.1 (0.9)

4. Secondary Outcome: Change in Physical Function as Measured Using the 6 Minute Walk Test
Description: Change in distance walked in six minutes from baseline
Time Frame: 0 weeks, 12 weeks
Population: Due to safety concerns during the COVID pandemic, the 6 Minute Walk Test was not administered to participants at all, so data from the 6 Minute Walk Test were not collected.
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Body Weight as Measured by the Aria Fitbit Scale
Description: Body weight in pounds.
Time Frame: 0 weeks, 12 weeks
Population: Participants who completed the study; data were not collected for one participant who completed.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 12
pounds
  0 weeks (baseline) | 216.1 (29.1)
  12 weeks | 215.4 (27.3)

6. Secondary Outcome: Change in Average Weekly Steps Measured Using Garmin Watch
Description: Average step counts using Garmin watch.
Time Frame: 0 weeks, 12 weeks
Population: Participants who completed the study; data were not collected for one participant who completed.
Measure: Mean (Standard Deviation); unit: steps per week
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 12
steps per week
  0 weeks (baseline) | 6204.8 (3802.1)
  12 weeks | 6365.0 (4109.8)

7. Secondary Outcome: Change in Total Calories Using 3-day Food Record (Participants Record Everything They Eat and Drink for Three Days)
Description: Average total calories consumed.
Time Frame: 0 weeks,12 weeks
Measure: Mean (Standard Deviation); unit: calories
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 11
calories
  Baseline | 1418.4 (364.7)
  12 weeks | 1525.8 (525.3)

8. Secondary Outcome: Change in Stress Using the Perceived Stress Scale
Description: Perceived Stress Scale is a 10-item stress assessment instrument. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Time Frame: 0 weeks, 12 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 13
score on a scale
  0 weeks (baseline) | 10.8 (5.2)
  12 weeks | 9.0 (4.3)

9. Secondary Outcome: Change in Self-reported Depression Using the Center for Epidemiologic Studies Depression Scale (CES-D)
Description: Score ranges from 0-60 with higher scores indicating greater depression symptoms.
Time Frame: 0 weeks, 12 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 13
score on a scale
  week 0 (baseline) | 11.3 (6.8)
  week 12 | 8.8 (7.0)

10. Secondary Outcome: Change in Mood Using the Profile of Mood States Questionnaire
Description: Change in mood from baseline, 6 and 12 weeks. Profile of Mood States is a psychological rating scale used to assess transient, distinct mood states that uses a five-point scale ranging from "not at all" to "extremely".
Time Frame: 0 weeks, 12 weeks
Population: To reduce participant burden during the COVID pandemic, this questionnaire was not administered to participants at all, so data from the Profile of Mood States (POMS) Questionnaire were not collected.
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 0

11. Secondary Outcome: Quality of Life Using the SF-36 Questionnaire - SF-36 Physical Functioning Scale
Description: Physical functioning scale of the SF-36 is a 10-items scale with a scores ranging from 0-100% where the higher score indicates greater physical functioning.
Time Frame: 0 weeks, 12 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 13
scores on a scale
  0 weeks (baseline) | 75.0 (18.7)
  12 weeks | 79.2 (20.6)

12. Secondary Outcome: Quality of Life Using the SF-36 Questionnaire - Role Limitations Due to Physical Health Scale
Description: Role limitations due to physical health scale of the SF-36 is a 4-items scale with a scores ranging from 0-100% where the higher score indicates less limitations due to physical health
Time Frame: 0 weeks, 12 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 13
scores on a scale
  0 weeks (baseline) | 59.6 (43.9)
  12 weeks | 75.0 (39.5)

13. Secondary Outcome: Quality of Life Using the SF-36 Questionnaire - Role Limitations Due to Emotional Problems Scale
Description: Role limitations due to emotional problems scale of the SF-36 is a 3-items scale with a scores ranging from 0-100% where the higher score indicates less limitations due to emotional health
Time Frame: 0 weeks, 12 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 13
scores on a scale
  0 weeks (baseline) | 66.7 (43.0)
  12 weeks | 64.1 (46.1)

14. Secondary Outcome: Quality of Life Using the SF-36 Questionnaire - Energy/Fatigue Scale
Description: Energy/fatigue scale of the SF-36 is a 4-items scale with a scores ranging from 0-100% where the higher score indicates less energy/fatigue
Time Frame: 0 weeks, 12 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 13
scores on a scale
  0 weeks (baseline) | 55.4 (21.6)
  12 weeks | 58.1 (20.5)

15. Secondary Outcome: Quality of Life Using the SF-36 Questionnaire - Emotional Well-Being Scale
Description: Emotional Well-Being scale of the SF-36 is a 5-items scale with a scores ranging from 0-100% where the higher score indicates greater emotional well-being
Time Frame: 0 weeks, 12 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 13
scores on a scale
  0 weeks (baseline) | 78.1 (13.6)
  12 weeks | 80.9 (10.6)

16. Secondary Outcome: Quality of Life Using the SF-36 Questionnaire - Social Functioning Scale
Description: Social Functioning scale of the SF-36 is a 2-items scale with a scores ranging from 0-100% where the higher score indicates greater social functioning.
Time Frame: 0 weeks, 12 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 13
scores on a scale
  0 weeks (baseline) | 82.7 (25.3)
  12 weeks | 83.7 (28.1)

17. Secondary Outcome: Quality of Life Using the SF-36 Questionnaire - Pain Scale
Description: Pain scale of the SF-36 is a 2-items scale with a scores ranging from 0-100% where the higher score indicates less pain.
Time Frame: 0 weeks, 12 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 13
scores on a scale
  0 weeks (baseline) | 68.5 (22.9)
  12 weeks | 75.2 (22.4)

18. Secondary Outcome: Quality of Life Using the SF-36 Questionnaire - General Health Scale
Description: General Health scale of the SF-36 is a 5-items scale with a scores ranging from 0-100% where the higher score indicates greater general health
Time Frame: 0 weeks, 12 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Legacy Intervention
Number analyzed (Participants) | 13
scores on a scale
  0 weeks (baseline) | 64.6 (15.5)
  12 weeks | 63.5 (18.0)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Legacy Intervention
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

LIMITATIONS AND CAVEATS:
Due to COVID restrictions, the research team had to minimize the number of in-person visits. Consequently, outcome measures data was only collected for baseline (0 weeks) and at 12 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT04490356/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT04490356/ICF_000.pdf